CLINICAL TRIAL: NCT05204836
Title: Altering Bone Microarchitecture and Mechanics by Off-label Pharmaceutical Intervention
Brief Title: Altering Bone Microarchitecture and Mechanics by Off-label Pharmaceutical Intervention Following an Acute Knee Injury
Acronym: ZAPOA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment stopped due to funding shortage. The scope of the original study increased beyond what had been budgeted in the grant that funded it, and follow-up funding attempts were not successful.
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB21-1109
Record Dates: First submitted 2021-12-21; First posted 2022-01-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries; Osteo Arthritis Knee
Keywords: acl tear; acl; acl rupture; acl injury; osteo arthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The cohort is randomized into a control and treatment group, where the treatment group receives a zoledronic acid injection within 6 weeks of ACL injury.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zoledronic Acid Injection (Experimental): Participants will receive 1 dose of 5 mg/100 mL intravenous zoledronic acid
  Interventions: Drug: Zoledronic Acid Injection
- Placebo (Placebo Comparator): Participants will receive 1 dose 100 ml Saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid Injection — 5 mg / 100 mL intravenous infusion
  Other Names: Taro-Zoledronic Acid; Dr. Reddy's Zoledronic Acid Injection
  Arms: Zoledronic Acid Injection
Drug: Placebo — 100 mL intravenous infusion
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if a zoledronic acid injection can alter the trajectory of joint degeneration following an acute anterior cruciate ligament (ACL) injury.

DETAILED DESCRIPTION:
After being informed about the study and potential risks and all participants giving written informed consent, this project will establish a cohort of young men and women who within six weeks have sustained an acute rupture of the ACL. The cohort is randomized into a control and treatment group, where the treatment group receives a zoledronic acid injection at baseline. The cohort will be followed radiographically with high resolution peripheral quantitative computed tomography (HR-pQCT), dual-energy computed tomography (DECT), digital radiography (X-Ray), bi-planar X-ray (EOS) and magnetic resonance imaging (MRI) for eighteen months to monitor the progression of joint changes and the effects of zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of an acute unilateral ACL tear (full-thickness, complete tear) will be recruited. This age range is chosen to ensure participants have fully developed adult bone structures and to exclude participants with menopause as this could affect study results.
* Participants with combined ligament deficiencies (posterior cruciate, medial and/or lateral collateral) or meniscal injury will be included. Participants must be able to fully extend the knee while supported at the time of the baseline measurement in order to conduct the HR-pQCT scan.
* Participants with a serum calcium level in the normal range (2.10-2.60 mmol/L) and a creatinine level above 59 (reported as eGFR) will be included.

Exclusion Criteria:

* Individuals with contraindications to zoledronic acid (see below)
* Prior knee ligament and/or meniscus tears, and/or intra-articular fractures.
* Females who are pregnant or planning pregnancy within a year will not be eligible. The research team will recommend participants who are planning to become pregnant within the next five years to withdraw their participation.
* Individuals with knees larger than the CT scanner's circular field of view.
* Individuals with a history of disease and/or treatment affecting bone turnover in the past 12 months.
* Individuals with injuries or implants that are not MRI-safe.

Zoledronic acid is contraindicated for:

* Patients who are hypersensitive to this drug or to any ingredient in the formulation, or to any bisphosphonates or component of the container.
* Severe renal impairment with creatinine clearance <35 mL/min and in those with evidence of acute renal impairment. For this study, participants with a creatinine clearance <50 mL/min may be excluded.
* Non-corrected hypocalcaemia at the time of infusion.
* Pregnant and nursing mothers.
* Patients who are already taking another bisphosphonate (ex. for osteoporosis).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Bone microarchitecture changes at 6 months as assessed by high resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline, 6 months
  To determine morphological parameters from HR-pQCT scans, the trabecular portion must be isolated from the cortical shell of the bone in order to analyse the components separately. This is accomplished with an already developed auto-segmentation algorithm. In addition, the raw HR-pQCT images must be converted to binary images, wherein each voxel (3D pixel) is either labelled 'bone' or 'not bone.' This segmentation is performed by an algorithm which applies either a Gaussian or Laplace-Hamming filter in addition to a threshold to the grey-scale images. The binary images can then be analysed and morphological parameters can be determined. The changes in bone microarchitecture will be assessed at 6 months in comparison to baseline.
Bone microarchitecture changes at 18 months as assessed by high resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline, 18 months
  To determine morphological parameters from HR-pQCT scans, the trabecular portion must be isolated from the cortical shell of the bone in order to analyse the components separately. This is accomplished with an already developed auto-segmentation algorithm. In addition, the raw HR-pQCT images must be converted to binary images, wherein each voxel (3D pixel) is either labelled 'bone' or 'not bone.' This segmentation is performed by an algorithm which applies either a Gaussian or Laplace-Hamming filter in addition to a threshold to the grey-scale images. The binary images can then be analysed and morphological parameters can be determined. The changes in bone microarchitecture will be assessed at 18 months in comparison to baseline.

SECONDARY OUTCOMES:
Bone marrow lesions (BML) and soft tissue injury changes at 2 months as assessed by Magnetic Resonance Imaging (MRI) | Baseline, 2 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using a threshold-based approach BMLs will be identified, and their location and volume will be recorded in cubic millimetres (mm^3). This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in the location and volume of the BMLs will be assessed at 2 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 2 months as assessed by Magnetic Resonance Imaging (MRI) | Baseline, 2 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular thickness which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular thickness will be assessed at 2 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 2 months as assessed by Magnetic Resonance Imaging (MRI) | Baseline, 2 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular separation which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular separation will be assessed at 2 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 2 months as assessed by Magnetic Resonance Imaging (MRI) | Baseline, 2 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of bone mineral density which will be recorded in milligrams of hydroxyapatite per cubic centimeter (mg HA/cm^3) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in bone mineral density will be assessed at 2 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 6 months as assessed by MRI | Baseline, 6 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using a threshold-based approach BMLs will be identified, and their location and volume will be recorded in cubic millimetres (mm^3). This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in the location and volume of the BMLs will be assessed at 6 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 6 months as assessed by MRI | Baseline, 6 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular thickness which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular thickness will be assessed at 6 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 6 months as assessed by MRI | Baseline, 6 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular separation which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular separation will be assessed at 6 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 6 months as assessed by MRI | Baseline, 6 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of bone mineral density which will be recorded in milligrams of hydroxyapatite per cubic centimeter (mg HA/cm^3) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in bone mineral density will be assessed at 6 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 18 months as assessed by MRI | Baseline, 18 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using a threshold-based approach BMLs will be identified, and their location and volume will be recorded in cubic millimetres (mm^3). This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in the location and volume of the BMLs will be assessed at 18 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 18 months as assessed by MRI | Baseline, 18 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular thickness which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular thickness will be assessed at 18 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 18 months as assessed by MRI | Baseline, 18 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of trabecular separation which will be recorded in millimeters (mm) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in trabecular separation will be assessed at 18 months comparison to baseline.
Bone marrow lesions (BML) and soft tissue injury changes at 18 months as assessed by MRI | Baseline, 18 months
  MRI data will be segmented to identify the bone surface in a similar fashion as described for HR-pQCT data. Using rigid body registration, the MRI data will be transformed to the HR-pQCT data, which allows for the analysis of bone mineral density which will be recorded in milligrams of hydroxyapatite per cubic centimeter (mg HA/cm^3) exclusively within the volume of BMLs. This analysis will be performed using custom algorithms in Python and the visualization toolkit. The changes in bone mineral density will be assessed at 18 months comparison to baseline.
Knee alignment as assessed by bi-planar x-ray | Baseline
  Joint alignment by bi-planar x-ray (EOS) In a standing position, the baseline study visit will capture the alignment of the tibia and femur bones bilaterally so that alignment of the knee joint can be assessed. This is a standard clinical imaging device, and the software for measurement of knee alignment is built into the system.
Patient reported outcomes using ACL Quality of Life Questionnaire - Baseline | Baseline
  Patient reported outcomes at baseline will be assessed using
  - ACL Quality of Life Questionnaire Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using ACL Quality of Life Questionnaire - 2 Months | 2 Months
  Patient reported outcomes at baseline will be assessed using
  - ACL Quality of Life Questionnaire Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using ACL Quality of Life Questionnaire - 6 Months | 6 Months
  Patient reported outcomes at baseline will be assessed using
  - ACL Quality of Life Questionnaire Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using ACL Quality of Life Questionnaire - 18 Months | 18 Months
  Patient reported outcomes at baseline will be assessed using
  - ACL Quality of Life Questionnaire Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using Knee injury and Osteoarthritis Outcome Score (KOOS) - Questionnaire - Baseline | Baseline
  Patient reported outcomes will be assessed using
  - Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Minimum Value: 1 (best outcome); Maximum Value: 5 (worse outcome)
Patient reported outcomes using Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire - 2 Months | 2 months
  Patient reported outcomes will be assessed using
  - Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Minimum Value: 1 (best outcome); Maximum Value: 5 (worse outcome)
Patient reported outcomes using Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire - 6 Months | 6 months
  Patient reported outcomes will be assessed using
  - Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Minimum Value: 1 (best outcome); Maximum Value: 5 (worse outcome)
Patient reported outcomes using Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire - 18 Months | 18 months
  Patient reported outcomes will be assessed using
  - Knee injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Minimum Value: 1 (best outcome); Maximum Value: 5 (worse outcome)
Patient reported outcomes using 36-Item Short Form Survey (SF-36) Questionnaire - Baseline | Baseline
  Patient reported outcomes will be assessed using
  - 36-Item Short Form Survey (SF-36) Questionnaire Questions 1, 2, 20, 22, 34, 36 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 3-12 - Minimum Value: 1 (worst outcome); Maximum Value: 3 (best outcome) Question 13-19 - Minimum Value: 1 (worst outcome); Maximum Value: 2 (best outcome) Questions 21, 23, 26, 27, 30 - Minimum Value: 1 (best outcome); Maximum Value: 6 (worst outcome) Questions 24, 25, 28, 29, 31 - Minimum Value: 1 (worst outcome); Maximum Value: 6 (best outcome) Questions 32, 33, 35 - Minimum Value: 1 (worst outcome); Maximum Value: 5 (best outcome)
Patient reported outcomes using 36-Item Short Form Survey (SF-36) Questionnaire - 2 months | 2 months
  Patient reported outcomes will be assessed using
  - 36-Item Short Form Survey (SF-36) Questionnaire Questions 1, 2, 20, 22, 34, 36 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 3-12 - Minimum Value: 1 (worst outcome); Maximum Value: 3 (best outcome) Question 13-19 - Minimum Value: 1 (worst outcome); Maximum Value: 2 (best outcome) Questions 21, 23, 26, 27, 30 - Minimum Value: 1 (best outcome); Maximum Value: 6 (worst outcome) Questions 24, 25, 28, 29, 31 - Minimum Value: 1 (worst outcome); Maximum Value: 6 (best outcome) Questions 32, 33, 35 - Minimum Value: 1 (worst outcome); Maximum Value: 5 (best outcome)
Patient reported outcomes using 36-Item Short Form Survey (SF-36) Questionnaire - 6 months | 6 months
  Patient reported outcomes will be assessed using
  - 36-Item Short Form Survey (SF-36) Questionnaire Questions 1, 2, 20, 22, 34, 36 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 3-12 - Minimum Value: 1 (worst outcome); Maximum Value: 3 (best outcome) Question 13-19 - Minimum Value: 1 (worst outcome); Maximum Value: 2 (best outcome) Questions 21, 23, 26, 27, 30 - Minimum Value: 1 (best outcome); Maximum Value: 6 (worst outcome) Questions 24, 25, 28, 29, 31 - Minimum Value: 1 (worst outcome); Maximum Value: 6 (best outcome) Questions 32, 33, 35 - Minimum Value: 1 (worst outcome); Maximum Value: 5 (best outcome)
Patient reported outcomes using 36-Item Short Form Survey (SF-36) Questionnaire - 18 months | 18 months
  Patient reported outcomes will be assessed using
  - 36-Item Short Form Survey (SF-36) Questionnaire Questions 1, 2, 20, 22, 34, 36 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 3-12 - Minimum Value: 1 (worst outcome); Maximum Value: 3 (best outcome) Question 13-19 - Minimum Value: 1 (worst outcome); Maximum Value: 2 (best outcome) Questions 21, 23, 26, 27, 30 - Minimum Value: 1 (best outcome); Maximum Value: 6 (worst outcome) Questions 24, 25, 28, 29, 31 - Minimum Value: 1 (worst outcome); Maximum Value: 6 (best outcome) Questions 32, 33, 35 - Minimum Value: 1 (worst outcome); Maximum Value: 5 (best outcome)
Patient reported outcomes using EQ-5D-5L Questionnaire - Baseline | Baseline
  Patient reported outcomes will be assessed using
  - EQ-5D-5L Questionnaire Questions 1-5 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 6 - Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using EQ-5D-5L Questionnaire - 2 months | 2 months
  Patient reported outcomes will be assessed using
  - EQ-5D-5L Questionnaire Questions 1-5 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 6 - Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using EQ-5D-5L Questionnaire - 6 months | 6 months
  Patient reported outcomes will be assessed using
  - EQ-5D-5L Questionnaire Questions 1-5 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 6 - Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes using EQ-5D-5L Questionnaire - 18 months | 18 months
  Patient reported outcomes will be assessed using
  - EQ-5D-5L Questionnaire Questions 1-5 - Minimum Value: 1 (best outcome); Maximum Value: 5 (worst outcome) Question 6 - Minimum Value: 0 (worst outcome); Maximum Value: 100 (best outcome)
Patient reported outcomes Health History Questionnaire (HHQ) - Baseline | Baseline
  Patient reported outcomes will be assessed using
  - Health History Questionnaire (HHQ) (No scale)
Patient reported outcomes Health History Questionnaire (HHQ) - 2 months | 2 months
  Patient reported outcomes will be assessed using
  - Health History Questionnaire (HHQ) (No scale)
Patient reported outcomes Health History Questionnaire (HHQ) - 6 months | 6 months
  Patient reported outcomes will be assessed using
  - Health History Questionnaire (HHQ) (No scale)
Patient reported outcomes Health History Questionnaire (HHQ) - 18 months | 18 months
  Patient reported outcomes will be assessed using
  - Health History Questionnaire (HHQ) (No scale)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Boyd, PhD, Principal Investigator — University of Calgary; Gregory Kline, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Dare D, Rodeo S. Mechanisms of post-traumatic osteoarthritis after ACL injury. Curr Rheumatol Rep. 2014 Oct;16(10):448. doi: 10.1007/s11926-014-0448-1. PMID 25182676
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Noyes FR, Bassett RW, Grood ES, Butler DL. Arthroscopy in acute traumatic hemarthrosis of the knee. Incidence of anterior cruciate tears and other injuries. J Bone Joint Surg Am. 1980 Jul;62(5):687-95, 757. PMID 7391091
- [Background] Speer KP, Spritzer CE, Bassett FH 3rd, Feagin JA Jr, Garrett WE Jr. Osseous injury associated with acute tears of the anterior cruciate ligament. Am J Sports Med. 1992 Jul-Aug;20(4):382-9. doi: 10.1177/036354659202000403. PMID 1415878
- [Background] Spindler KP, Schils JP, Bergfeld JA, Andrish JT, Weiker GG, Anderson TE, Piraino DW, Richmond BJ, Medendorp SV. Prospective study of osseous, articular, and meniscal lesions in recent anterior cruciate ligament tears by magnetic resonance imaging and arthroscopy. Am J Sports Med. 1993 Jul-Aug;21(4):551-7. doi: 10.1177/036354659302100412. PMID 8368416
- [Background] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Background] Poulsen E, Goncalves GH, Bricca A, Roos EM, Thorlund JB, Juhl CB. Knee osteoarthritis risk is increased 4-6 fold after knee injury - a systematic review and meta-analysis. Br J Sports Med. 2019 Dec;53(23):1454-1463. doi: 10.1136/bjsports-2018-100022. Epub 2019 May 9. PMID 31072840
- [Background] Buckwalter JA. Articular cartilage injuries. Clin Orthop Relat Res. 2002 Sep;(402):21-37. doi: 10.1097/00003086-200209000-00004. PMID 12218470
- [Background] Claes S, Hermie L, Verdonk R, Bellemans J, Verdonk P. Is osteoarthritis an inevitable consequence of anterior cruciate ligament reconstruction? A meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):1967-76. doi: 10.1007/s00167-012-2251-8. Epub 2012 Oct 26. PMID 23100047
- [Background] Huetink K, Nelissen RG, Watt I, van Erkel AR, Bloem JL. Localized development of knee osteoarthritis can be predicted from MR imaging findings a decade earlier. Radiology. 2010 Aug;256(2):536-46. doi: 10.1148/radiol.10090683. Epub 2010 Jun 29. PMID 20587644
- [Background] Meunier A, Odensten M, Good L. Long-term results after primary repair or non-surgical treatment of anterior cruciate ligament rupture: a randomized study with a 15-year follow-up. Scand J Med Sci Sports. 2007 Jun;17(3):230-7. doi: 10.1111/j.1600-0838.2006.00547.x. PMID 17501866
- [Background] Hunter DJ, Guermazi A, Lo GH, Grainger AJ, Conaghan PG, Boudreau RM, Roemer FW. Evolution of semi-quantitative whole joint assessment of knee OA: MOAKS (MRI Osteoarthritis Knee Score). Osteoarthritis Cartilage. 2011 Aug;19(8):990-1002. doi: 10.1016/j.joca.2011.05.004. Epub 2011 May 23. PMID 21645627
- [Background] Bhatla JL, Kroker A, Manske SL, Emery CA, Boyd SK. Differences in subchondral bone plate and cartilage thickness between women with anterior cruciate ligament reconstructions and uninjured controls. Osteoarthritis Cartilage. 2018 Jul;26(7):929-939. doi: 10.1016/j.joca.2018.04.006. Epub 2018 Apr 17. PMID 29678623
- [Background] Kroker A, Manske SL, Mohtadi N, Boyd SK. A study of the relationship between meniscal injury and bone microarchitecture in ACL reconstructed knees. Knee. 2018 Oct;25(5):746-756. doi: 10.1016/j.knee.2018.07.004. Epub 2018 Aug 13. PMID 30115589
- [Background] Michalak GJ, Walker R, Boyd SK. Concurrent Assessment of Cartilage Morphology and Bone Microarchitecture in the Human Knee Using Contrast-Enhanced HR-pQCT Imaging. J Clin Densitom. 2019 Jan-Mar;22(1):74-85. doi: 10.1016/j.jocd.2018.07.002. Epub 2018 Jul 19. PMID 30120027
- [Background] Kroker A, Bhatla JL, Emery CA, Manske SL, Boyd SK. Subchondral bone microarchitecture in ACL reconstructed knees of young women: A comparison with contralateral and uninjured control knees. Bone. 2018 Jun;111:1-8. doi: 10.1016/j.bone.2018.03.006. Epub 2018 Mar 8. PMID 29526780
- [Background] Kroker A, Besler BA, Bhatla JL, Shtil M, Salat P, Mohtadi N, Walker RE, Manske SL, Boyd SK. Longitudinal Effects of Acute Anterior Cruciate Ligament Tears on Peri-Articular Bone in Human Knees Within the First Year of Injury. J Orthop Res. 2019 Nov;37(11):2325-2336. doi: 10.1002/jor.24410. Epub 2019 Jul 23. PMID 31283044
- [Background] She G, Zhou Z, Zha Z, Wang F, Pan X. Protective effect of zoledronic acid on articular cartilage and subchondral bone of rabbits with experimental knee osteoarthritis. Exp Ther Med. 2017 Nov;14(5):4901-4909. doi: 10.3892/etm.2017.5135. Epub 2017 Sep 19. PMID 29201194
- [Background] Spector TD, Conaghan PG, Buckland-Wright JC, Garnero P, Cline GA, Beary JF, Valent DJ, Meyer JM. Effect of risedronate on joint structure and symptoms of knee osteoarthritis: results of the BRISK randomized, controlled trial [ISRCTN01928173]. Arthritis Res Ther. 2005;7(3):R625-33. doi: 10.1186/ar1716. Epub 2005 Mar 24. PMID 15899049
- [Background] Bingham CO 3rd, Buckland-Wright JC, Garnero P, Cohen SB, Dougados M, Adami S, Clauw DJ, Spector TD, Pelletier JP, Raynauld JP, Strand V, Simon LS, Meyer JM, Cline GA, Beary JF. Risedronate decreases biochemical markers of cartilage degradation but does not decrease symptoms or slow radiographic progression in patients with medial compartment osteoarthritis of the knee: results of the two-year multinational knee osteoarthritis structural arthritis study. Arthritis Rheum. 2006 Nov;54(11):3494-507. doi: 10.1002/art.22160. PMID 17075851
- [Background] Adami S, Pavelka K, Cline GA, Hosterman MA, Barton IP, Cohen SB, Bensen WG. Upper gastrointestinal tract safety of daily oral risedronate in patients taking NSAIDs: a randomized, double-blind, placebo-controlled trial. Mayo Clin Proc. 2005 Oct;80(10):1278-85. doi: 10.4065/80.10.1278. PMID 16212139
- [Background] Laslett LL, Dore DA, Quinn SJ, Boon P, Ryan E, Winzenberg TM, Jones G. Zoledronic acid reduces knee pain and bone marrow lesions over 1 year: a randomised controlled trial. Ann Rheum Dis. 2012 Aug;71(8):1322-8. doi: 10.1136/annrheumdis-2011-200970. Epub 2012 Feb 21. PMID 22355040
- [Background] Rossini M, Adami S, Fracassi E, Viapiana O, Orsolini G, Povino MR, Idolazzi L, Gatti D. Effects of intra-articular clodronate in the treatment of knee osteoarthritis: results of a double-blind, randomized placebo-controlled trial. Rheumatol Int. 2015 Feb;35(2):255-63. doi: 10.1007/s00296-014-3100-5. Epub 2014 Aug 1. PMID 25080876
- [Background] Varenna M, Zucchi F, Failoni S, Becciolini A, Berruto M. Intravenous neridronate in the treatment of acute painful knee osteoarthritis: a randomized controlled study. Rheumatology (Oxford). 2015 Oct;54(10):1826-32. doi: 10.1093/rheumatology/kev123. Epub 2015 May 20. PMID 25998450
- [Background] Vaysbrot EE, Osani MC, Musetti MC, McAlindon TE, Bannuru RR. Are bisphosphonates efficacious in knee osteoarthritis? A meta-analysis of randomized controlled trials. Osteoarthritis Cartilage. 2018 Feb;26(2):154-164. doi: 10.1016/j.joca.2017.11.013. Epub 2017 Dec 6. PMID 29222056
- [Background] Kuttapitiya A, Assi L, Laing K, Hing C, Mitchell P, Whitley G, Harrison A, Howe FA, Ejindu V, Heron C, Sofat N. Microarray analysis of bone marrow lesions in osteoarthritis demonstrates upregulation of genes implicated in osteochondral turnover, neurogenesis and inflammation. Ann Rheum Dis. 2017 Oct;76(10):1764-1773. doi: 10.1136/annrheumdis-2017-211396. Epub 2017 Jul 13. PMID 28705915
- [Background] Cai G, Aitken D, Laslett LL, Pelletier JP, Martel-Pelletier J, Hill C, March L, Wluka AE, Wang Y, Antony B, Blizzard L, Winzenberg T, Cicuttini F, Jones G. Effect of Intravenous Zoledronic Acid on Tibiofemoral Cartilage Volume Among Patients With Knee Osteoarthritis With Bone Marrow Lesions: A Randomized Clinical Trial. JAMA. 2020 Apr 21;323(15):1456-1466. doi: 10.1001/jama.2020.2938. PMID 32315057
- [Background] Aitken D, Laslett LL, Cai G, Hill C, March L, Wluka AE, Wang Y, Blizzard L, Cicuttini F, Jones G. A protocol for a multicentre, randomised, double-blind, placebo-controlled trial to compare the effect of annual infusions of zoledronic acid to placebo on knee structural change and knee pain over 24 months in knee osteoarthritis patients - ZAP2. BMC Musculoskelet Disord. 2018 Jul 18;19(1):217. doi: 10.1186/s12891-018-2143-2. PMID 30021646
- [Background] Lohmander LS, Ostenberg A, Englund M, Roos H. High prevalence of knee osteoarthritis, pain, and functional limitations in female soccer players twelve years after anterior cruciate ligament injury. Arthritis Rheum. 2004 Oct;50(10):3145-52. doi: 10.1002/art.20589. PMID 15476248
- [Background] Davis AM, Kennedy D, Wong R, Robarts S, Skou ST, McGlasson R, Li LC, Roos E. Cross-cultural adaptation and implementation of Good Life with osteoarthritis in Denmark (GLA:D): group education and exercise for hip and knee osteoarthritis is feasible in Canada. Osteoarthritis Cartilage. 2018 Feb;26(2):211-219. doi: 10.1016/j.joca.2017.11.005. Epub 2017 Nov 13. PMID 29146385
- [Background] Maetzel A, Li LC, Pencharz J, Tomlinson G, Bombardier C; Community Hypertension and Arthritis Project Study Team. The economic burden associated with osteoarthritis, rheumatoid arthritis, and hypertension: a comparative study. Ann Rheum Dis. 2004 Apr;63(4):395-401. doi: 10.1136/ard.2003.006031. PMID 15020333
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Burt LA, Liang Z, Sajobi TT, Hanley DA, Boyd SK. Sex- and Site-Specific Normative Data Curves for HR-pQCT. J Bone Miner Res. 2016 Nov;31(11):2041-2047. doi: 10.1002/jbmr.2873. Epub 2016 Jun 9. PMID 27192388
- [Background] Campbell GM, Buie HR, Boyd SK. Signs of irreversible architectural changes occur early in the development of experimental osteoporosis as assessed by in vivo micro-CT. Osteoporos Int. 2008 Oct;19(10):1409-19. doi: 10.1007/s00198-008-0581-7. Epub 2008 Mar 29. PMID 18373058
- [Background] Whittier DE, Boyd SK, Burghardt AJ, Paccou J, Ghasem-Zadeh A, Chapurlat R, Engelke K, Bouxsein ML. Guidelines for the assessment of bone density and microarchitecture in vivo using high-resolution peripheral quantitative computed tomography. Osteoporos Int. 2020 Sep;31(9):1607-1627. doi: 10.1007/s00198-020-05438-5. Epub 2020 May 26. PMID 32458029
- [Background] Mattap SM, Aitken D, Wills K, Laslett L, Ding C, Pelletier JP, Martel-Pelletier J, Graves SE, Lorimer M, Cicuttini F, Jones G. How Do MRI-Detected Subchondral Bone Marrow Lesions (BMLs) on Two Different MRI Sequences Correlate with Clinically Important Outcomes? Calcif Tissue Int. 2018 Aug;103(2):131-143. doi: 10.1007/s00223-018-0402-8. Epub 2018 Feb 13. PMID 29441423
- [Background] Guermazi A, Eckstein F, Hellio Le Graverand-Gastineau MP, Conaghan PG, Burstein D, Keen H, Roemer FW. Osteoarthritis: current role of imaging. Med Clin North Am. 2009 Jan;93(1):101-26, xi. doi: 10.1016/j.mcna.2008.08.003. PMID 19059024
- [Background] Kroker A, Zhu Y, Manske SL, Barber R, Mohtadi N, Boyd SK. Quantitative in vivo assessment of bone microarchitecture in the human knee using HR-pQCT. Bone. 2017 Apr;97:43-48. doi: 10.1016/j.bone.2016.12.015. Epub 2016 Dec 27. PMID 28039095
- [Background] Compston J. Pathophysiology of atypical femoral fractures and osteonecrosis of the jaw. Osteoporos Int. 2011 Dec;22(12):2951-61. doi: 10.1007/s00198-011-1804-x. Epub 2011 Oct 14. PMID 21997225
- [Background] Mohtadi N. Development and validation of the quality of life outcome measure (questionnaire) for chronic anterior cruciate ligament deficiency. Am J Sports Med. 1998 May-Jun;26(3):350-9. doi: 10.1177/03635465980260030201. PMID 9617395
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Buie HR, Campbell GM, Klinck RJ, MacNeil JA, Boyd SK. Automatic segmentation of cortical and trabecular compartments based on a dual threshold technique for in vivo micro-CT bone analysis. Bone. 2007 Oct;41(4):505-15. doi: 10.1016/j.bone.2007.07.007. Epub 2007 Jul 18. PMID 17693147
- [Background] Kemp TD, de Bakker CMJ, Gabel L, Hanley DA, Billington EO, Burt LA, Boyd SK. Longitudinal bone microarchitectural changes are best detected using image registration. Osteoporos Int. 2020 Oct;31(10):1995-2005. doi: 10.1007/s00198-020-05449-2. Epub 2020 May 19. PMID 32430614
- [Background] Ellouz R, Chapurlat R, van Rietbergen B, Christen P, Pialat JB, Boutroy S. Challenges in longitudinal measurements with HR-pQCT: evaluation of a 3D registration method to improve bone microarchitecture and strength measurement reproducibility. Bone. 2014 Jun;63:147-57. doi: 10.1016/j.bone.2014.03.001. Epub 2014 Mar 12. PMID 24614646
- [Background] Arias-Moreno AJ, Hosseini HS, Bevers M, Ito K, Zysset P, van Rietbergen B. Validation of distal radius failure load predictions by homogenized- and micro-finite element analyses based on second-generation high-resolution peripheral quantitative CT images. Osteoporos Int. 2019 Jul;30(7):1433-1443. doi: 10.1007/s00198-019-04935-6. Epub 2019 Apr 17. PMID 30997546